CLINICAL TRIAL: NCT04794998
Title: A Simple Approach to Treat COVID-19 Patients at Home: Does it Reduce Recovery Time? A Retrospective Observational Matched-cohort Study
Brief Title: A Simple Approach to Treat COVID-19 Patients at Home.
Acronym: COVER
Status: Completed | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: COVER
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: COVID 19
Keywords: COVID-19 treatment
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- "Recommended schedule" cohort: COVID-19 patients who have applied the proposed treatment recommendation algorithm at the onset of or within few days from the beginning of symptoms.
  Interventions: Drug: Recommended treatment schedule
- "control" cohort: COVID-19 patients enrolled in the ORIGIN study of the Istituto di Ricerche Farmacologiche Mario Negri IRCCS, and treated at home by their family doctors with drug regimens other than those proposed in the recommendations
  Interventions: Drug: Control treatment schedule

INTERVENTIONS:
Drug: Recommended treatment schedule — Relatively selective Cox-2 inhibitors, Corticosteroids (Dexamethasone), Anticoagulants (LMW heparin), Gentle Oxygen therapy
  Groups: "Recommended schedule" cohort
Drug: Control treatment schedule — Treatment regimens different from the recommended one according to family phisicians personal practice.
  Groups: "control" cohort

SUMMARY:
The newly recognised disease COVID-19 is caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), which by early December 2019 had spread from China to the rest of the world, especially Europe, the United States, Latin America, and India, with over 86 million confirmed cases and over 1.870.000 deaths (5th January, 2021). The clinical spectrum of SARSCoV- 2 infection is wide, encompassing asymptomatic infection, mild upper respiratory tract illness, and severe viral pneumonia with respiratory failure and even death.

According to retrospective data from China regarding 1099 patients with laboratory-confirmed COVID-19, at the time of admission to hospital, the most common symptoms were cough (67.8%), fever (43%), and fatigue (38.1%), and less frequently myalgia/arthralgia (14.9%), a sore throat (13.9%) and headache (13.6), while nausea or vomiting (5.0%) and diarrhoea (3.8%) were uncommon. Similar clinical characteristics are also encountered in European and US COVID-19 patients.

Given the rising global death toll associated with the pandemic, in the past few months we have witnessed a race to find drug/biological treatments to save the lives of hospitalized, severely ill patients, as well as to develop vaccines. To this end, randomized clinical trials are underway to test experimental drug candidates, or repurposed medicines. At this time, it is crucial to focus on primary care physicians and initial mild symptoms at home in COVID-19 patients.

Recently recommendations have been produced to treat this illness at home based on the pathophysiologic and the pharmacologic rationale and the available clinical evidence of efficacy in COVID-19 patients, including results of published clinical trials, for each of the recommended class of drugs. These recommendations have taken advantage from the long term experience of an infection disease specialist and other clinicians of Bergamo Hospital, who used their know-how and sound judgment to treat COVID-19 patients at home.

Because the common early mild symptoms of COVID-19 highlight a systemic inflammatory process, there is the recommendation of using anti-inflammatory agents to limit excessive host inflammatory responses to the viral infection, including non-steroidal anti-inflammatory drugs and corticosteroids.

Moreover, COVID-19 is a particularly debilitating illness, and, apart from causing patients to be bedridden, there is evidence that in SARS-CoV-2 infection, dysregulation of the coagulation cascade and fibrinolytic system occur. Therefore, COVID-19 patients are exposed to the risk of thromboembolic events, independently of age, and anticoagulant prophylaxis is recommended, unless contraindicated.

Comparative analysis of patient cohorts with long-enough follow-up in everyday clinical practice may offer a good alternative to randomized clinical trials to evaluate effectiveness of novel therapies. Thus, we will use this approach in an observational retrospective matched-cohort study to compare a cohort of COVID-19 patients treated at home by their family phisicians according to the proposed recommendations with another cohort of similar patients treated with other therapeutic regimens.

Our working hypothesis is that following the recommendations the inflammatory processes and thus symptoms resolve faster than with other therapeutic approaches, while safe achieving similar rates of complete remission of the illness.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult (≥18 years old)
* Subjects with early mild symptoms of COVID-19, without waiting results of a nasopharyngeal swab, if any
* Informed consent

Exclusion Criteria:

* Subjects who require immediate hospital admission because severe COVID-19 symptoms at onset according to family doctor opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients treated at home by their family doctors according to the proposed recommendations from May 2020 to November 2020. It will include all available family physicians who have followed these recommendations and expressed interest in the study.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Time to complete remission | From beginning the proposed recommended treatments or other therapeutic regimens to resolution of major symptoms, assessed up to 20 days.
  "Complete remission" is defined as complete recovery from major symptoms, ie no fever, SpO2 >94% and/or no dyspnea, no cough, no rhinitis, no pain (myalgia, arthralgia, chest pain, headache, sore throat), no vertigo, no nausea, vomiting or diarrhoea, no sicca syndrome or red eyes.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Reserach Center for Rare Diseases "Aldo e Cele Daccò", Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: Undecided